CLINICAL TRIAL: NCT03182036
Title: Portable Oxygen Concentrator Signal Capture Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: St George Hospital, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR110517
Record Dates: First submitted 2017-05-16; First posted 2017-06-09 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study group (Experimental): Portable pulsed oxygen
  Interventions: Device: Portable pulsed oxygen

INTERVENTIONS:
Device: Portable pulsed oxygen — Hypoxemic patients will use portable pulsed oxygen at rest, and while performing a six-minute walk test.

SUMMARY:
The main purpose of this study is to learn how patients breathe on portable oxygen concentrators (POCs), and to get feedback from patients using POCs.

DETAILED DESCRIPTION:
This study aims to examine patient oxygenation levels and markers of exertion (e.g. breath rate, heart rate and breath pattern) while using a portable oxygen concentrator, with the aim to understand exercise desaturation in hypoxemic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to give written informed consent
* Patient can read and comprehend English
* Patient is ≥ 18 years of age
* Patient has moderate to severe hypoxaemia (SpO2 ≤ 92%) at rest
* Patient reports shortness of breath on exertion

Exclusion Criteria:

* Patient has musculoskeletal impairment, or other impairment that may be the limiting factor in 6MWT
* Patient has a history of a psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study
* Patient has acute coronary syndrome, acute myo- or pericarditis, acute lung embolism, pulmonary infarction, acute uncontrolled heart insufficiency
* Patient shows signs of acute exacerbation of underlying lung condition
* Patient is deemed to be unsuitable for inclusion in the opinion of the researcher, including for the following reasons:
* they do not comprehend English
* they are unable to provide written informed consent
* they are physically unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Oxygenation | 20 minutes
  SpO2 during rest and exercise using portable pulsed oxygen therapy

SECONDARY OUTCOMES:
Heart rate | 20 minutes
  Heart rate during rest and exercise using portable pulsed oxygen therapy
Nasal cannula pressure | 20 minutes
  Nasal cannula pressure during rest and exercise using portable pulsed oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Dickens, PhD, Study Director — ResMed; Peter Wlodarczyk, BEng, Study Director — ResMed
Locations (1):
- St George Hospital, Kogarah, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No